CLINICAL TRIAL: NCT02275364
Title: A Magnetic Resonance Imaging Study of Nasal Strips in Subjects With Nasal Congestion
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Study of Nasal Strips in Nasal Congestion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 202178
Record Dates: First submitted 2014-05-22; First posted 2014-10-27 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Nasal Congestion
MeSH Terms: conditions — Nasal Obstruction | interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test nasal strip (Experimental): Marketed Nasal Strip to be applied for up to two hours, and during the third scanning session for approximately 20 minutes.
  Interventions: Device: Test strip; Other: Nasal spray
- Placebo nasal strip (Placebo Comparator): Placebo nasal strip to be applied for up to two hours in either of the first two scans only.
  Interventions: Device: Placebo strip; Other: Nasal spray

INTERVENTIONS:
Device: Test strip — Class I device for the application to the nose to facilitate better air flow through the nose
  Arms: Test nasal strip
Device: Placebo strip — Placebo strip
  Arms: Placebo nasal strip
Other: Nasal spray — Nasal decongestant to be used on a single occasion (one spray per nostril), 20 minutes prior to commencing the third MRI scanning sessions.

SUMMARY:
The aim of the study is to evaluate the effect of the nasal strip (relative to the placebo strip) on the nasal passages using anatomical MRI scans and to demonstrate the effect of the strip on breathing correlated cortical activity, using interoceptive fMRI task and analysis techniques derived from physiological data collected during scanning.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a self-rating of at least 3 to 8 for nasal congestion on the numerical rating scale
* Participants with a nasal congestion frequency score of 1, 2, 3 or 4.

Exclusion Criteria:

* Evidence of obstructive nasal polyps, nasal tract structural malformations, visible open sores, sunburn, irritation, eczema or chronic skin condition on the face or nose
* Use of any medications like nasal decongestant, alpha adrenergic drugs, glucocorticoids and any current treatment which in the opinion of the investigator will affect nasal congestion
* Known or suspected intolerance or hypersensitivity to the study materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2013-10-30 (Actual); Study Completion 2013-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Imanova Centre for Imaging Sciences, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a clinical site in London.
Pre-assignment Details: A total of 35 participants were screened of which 28 were randomized in the study. Five of these did not meet study criteria, 1 had a protocol violation and 1 additional participant had other reason to leave the study, prior to be randomized.
Groups:
- Sequence 1: In the sequence 1 of the crossover part of the study, participants were randomized to receive placebo strip first (period 1) followed by marketed strip (period 2). The placebo strip was applied for up to two hours for the first scanning sessions, and then removed and the marketed strip applied for the second scanning session. The strip was removed and participants applied the nasal spray (period 3) and then after approximately 30 minutes, applied the marketed nasal strip for the third scanning session (period 4). There was no washout for period 3, as treatment B i.e. marketed nasal strip, was added in period 4 to the nasal decongestant spray that was applied in period 3
- Sequence 2: In the sequence 1 of the crossover part of the study, participants were randomized to receive marketed strip first (period 1) followed by marketed strip (period 2). The marketed strip was applied for up to two hours for the first scanning sessions, and then removed and the placebo strip applied for the second scanning session. The strip was removed and participants applied the nasal spray (period 3) and then after approximately 30 minutes, applied the marketed nasal strip for the third scanning session (period 4). There was no washout for period 3, as treatment B i.e. marketed nasal strip, was added in period 4 to the nasal decongestant spray that was applied in period 3
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 14 | 14
Completed | 12 | 14
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other reason | 1 | 0
Period: Washout Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Participants were randomized to receive either Marketed Nasal Strip or Placebo Nasal Strip (to be applied for up to two hours in either of the first two scans only). During the third scanning session, Marketed Nasal Strip was applied for approximately 20 minutes after administration of a Marketed Decongestant.
Arm/Group | Overall
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Anatomical Measures : Cross Sectional Area
Description: Determination of cross sectional area derived from examination of the nasal passages and sinuses using T1 weighted MRI scans.
Time Frame: Upto 2.5 hours
Population: Per-Protocol (PP) Population: Participants successfully completing all conditions of the experiment on single visit day except whose data didn't meet quality standards (problems with devices/software or participant (excessive head-motion during fMRI, inadequate performance of experimental tasks). Data of 7 participants didn't meet the standards.
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Test Nasal Strip: Marketed Nasal Strip to be applied for up to two hours, in either of the first two sessions
- Decongestant: A Nasal Decongestant was administered (one spray per nostril) by the participants 20 mins (+/- 5 mins) prior to the third MRI scanning session.
- Test Nasal Strip Plus Decongestant: Marketed Nasal Strip to be applied during the third scanning session for approximately 20 minutes, after administration of a Marketed Decongestant.
Arm/Group | Test Nasal Strip | Placebo Nasal Strip | Decongestant | Test Nasal Strip Plus Decongestant
Number analyzed (Participants) | 21 | 21 | 21 | 21
mm^2 | 133.22 (28.946) | 116.88 (31.468) | 156.48 (29.103) | 176.12 (29.370)
Statistical Analysis 1: Comparison: Test Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p < 0.0001, ANOVA — Obtained from ANOVA model with Treatment and Period as fixed effects and subject as a random effect; Adjusted Mean Difference = 15.28, 95% CI 2-sided [12.32 to 18.25] — Adjusted Mean Difference is the treatment difference defined as the Adjusted Mean of Test Nasal Strip minus Adjusted Mean of Placebo Strip

2. Primary Outcome: Functional Brain Activity: Blood Oxygen Level Dependent- Interoceptive Attention Task
Description: Regional measures of functional brain activity to be derived from a breathing-related interoceptive task. This outcome measure was pre-specified to analyze effect on nasal strips on the functional brain activity without the use of nasal decongestant.
Time Frame: Upto 2.5 hours
Population: Decongestant and Test Nasal Strip Plus Decongestant groups were not included in this outcome measure as it was pre-specified to analyze effect on nasal strips on the brain activity without the use of nasal decongestant
Measure: Mean (Standard Deviation); unit: % Signal
Groups:
- Marketed Nasal Strip: Marketed Nasal Strip to be applied for up to two hours, and during the third scanning session for approximately 20 minutes.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip
Number analyzed (Participants) | 25 | 25
% Signal | 7.39 (9.858) | 7.92 (8.246)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.7366, ANCOVA — Obtained from ANOVA with treatment, period and region of interest as fixed effects and subject as a random effect; Adjusted Mean Difference = -0.93, 95% CI 2-sided [-6.43 to 4.57] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Anatomical Measure: Volume (Single Volume Reading)
Description: Determination of single volume reading derived from examination of the nasal passages and sinuses, during the MRI.
Time Frame: Upto 2.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Marketed Nasal Strip Plus Decongestant: Marketed Nasal Strip to be applied during the third scanning session for approximately 20 minutes, after administration of a Marketed Decongestant.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Decongestant | Marketed Nasal Strip Plus Decongestant
Number analyzed (Participants) | 21 | 21 | 21 | 21
mm^3 | 13407.42 (3199.592) | 11732.85 (3254.077) | 15770.79 (3596.181) | 17680.49 (3691.798)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.0004, ANOVA — Obtained from ANOVA model with Treatment and Period as fixed effects and subject as a random effect; Adjusted Mean Difference = 1533.74, 95% CI 2-sided [794.16 to 2273.32] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cerebral Blood Flow (CBF)
Description: CBF was derived from Arterial-Spin Labelling (ASL) scans. ASL data were analysed using custom Matlab code, which fits a CBF model to the raw perfusion data, in order to derive quantitative estimates of CBF in units of ml/100g/minute. The computed CBF maps were co-registered to the subject's whole-brain T1-weighted anatomical scan (from the first scan session) in order to spatially divide the data into anatomical Regions of Interest (ROIs). The anatomical ROIs were themselves defined by nonlinear warping of a standard cytoarchitectonic atlas into the space of the subject's T1 anatomical scan, using the FMRIB Software Library tool FNIRT. CBF data were extracted for a subset of these anatomical ROIs.
Time Frame: Upto 2.5 hours
Population: Decongestant and Test Nasal Strip Plus Decongestant groups were not evaluated in this outcome measure as it was pre-specified to to analyze effect of nasal strips on the cerebral blood without the use of nasal decongestant.
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip
Number analyzed (Participants) | 21 | 21
ml/100g/min | 85.80 (23.351) | 86.25 (20.079)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.7278, ANOVA — Obtained from ANOVA model with Treatment and Period as fixed effects and subject as a random effect; Adjusted Mean Difference = -0.46, 95% CI 2-sided [-3.06 to 2.14] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Anatomical Measures: Volume (Multiple Volume Reading)
Description: Determination of averaged volume reading during the MRI (Average of 8 sub-regions)
Time Frame: Upto 2.5 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Decongestant: A marketed nasal decongestant was administered (one spray per nostril) by the participants 20 mins (+/- 5 mins) prior to the third MRI scanning session.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Decongestant | Marketed Nasal Strip Plus Decongestant
Number analyzed (Participants) | 21 | 21 | 21 | 21
mm^3 | 1675.93 (399.949) | 1466.61 (406.760) | 1971.35 (449.523) | 2210.06 (461.475)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.1639, ANCOVA — Obtained from ANOVA model with Treatment and Period as fixed effects and subject as a random effect; Adjusted Mean Difference = 191.72, 95% CI 2-sided [-78.62 to 462.06] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Functional Measure: Blood Oxygen Level Dependent- Interoceptive Attention Task (Psychophysiological Interactive Analysis)
Description: Regional measures of functional brain activity were to be derived from a breathing-related interoceptive task.
Time Frame: Upto 2.5 hours
Population: Decongestant and Test Nasal Strip Plus Decongestant groups were not included in this outcome measure as it was pre-specified to evaluate the effect on nasal strips on the measure of brain activity without the use of nasal decongestant.
Measure: Mean (Standard Deviation); unit: % signal change
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip
Number analyzed (Participants) | 25 | 25
% signal change | 0.13 (0.123) | 0.12 (0.161)
Statistical Analysis 1: Comparison: Marketed Nasal Strip vs Placebo Nasal Strip; Test type: Superiority or Other; p = 0.4621, ANOVA — Obtained from ANOVA with treatment, period and region of interest as fixed effects and subject as a random effect; Adjusted Mean Difference = 0.02, 95% CI 2-sided [-0.03 to 0.07] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Breathing-related Cortical Activity (Blood Oxygen Level Dependent- Resting State)
Description: Regional measures of breathing-related cortical activity were derived by determining Functional Connectivity and Event-related percentage signal change.
  Functional connectivity analyzes of fMRI data where spontaneous (i.e. while the participant is at rest) signal changes in one brain region are regressed against other regions, to identify regions sharing similar functional properties.
  Event-related functional magnetic resonance imaging (efMRI) detects changes in the BOLD hemodynamic response to neural activity associated with certain event. In this case, the events were pre-defined by collecting additional data during the scan; participant respiration was determined using a simple pressure-sensitive respiration belt. Events time-locked to peak inspiration and expiration were defined separately, and regressed against brain activity, showing brain regions that were more or less active during each event type.
Time Frame: Upto 2.5 hours
Population: Decongestant and Test Nasal Strip Plus Decongestant groups were not included in this outcome measure as it was prespecified to evaluate the effect on nasal strips on the breathing related brain activity without the use of nasal decongestant
Measure: Mean (Standard Deviation); unit: % signal change
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip
Number analyzed (Participants) | 25 | 25
% signal change
  Functional Connectivity (% signal change) | 0.42 (0.261) | 0.33 (0.249)
  Event-related (% signal change) | 27.57 (40.038) | 10.80 (43.793)

8. Secondary Outcome: Verbal Numerical Response (VNR): Change From Baseline to Immediately After Strip Application and 30 Minutes Post Application
Description: Participants provided their response for VNR on a scale of 0 to 10 (0 = Breathe Freely and 10 = Totally Blocked) how easy it was to breathe through nose at a given time.
Time Frame: Upto 30 minutes
Population: Per-Protocol (PP) Population: Participants successfully completing all conditions of the experiment on single visit day except whose data didn't meet quality standards (problems with devices/software or participant (excessive head-motion during fMRI, inadequate performance of experimental tasks). Data of 2 participants didn't meet the standards.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo Strip: Placebo nasal strip to be applied for up to two hours in either of the first two scans only.
Arm/Group | Test Nasal Strip | Placebo Strip
Number analyzed (Participants) | 26 | 26
Units on a scale
  Immediate Change from Baseline (Units on a scale) | -0.46 (1.067) | -0.07 (0.900)
  30 minutes Change from Baseline (Units on a scale) | -1.00 (1.296) | -0.42 (1.629)

9. Secondary Outcome: VNR: Change From Baseline to 20 Minutes After Decongestant Administration, and Post Application of the Marketed Nasal Strip After Decongestant Administration
Description: as for outcome 8
Time Frame: Upto 2 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Marketed Nasal Strip Plus Decongestant
Number analyzed (Participants) | 26
Units on a scale
  Change from baseline post-decongestant use | -1.35 (1.522)
  Change from baseline (Nasal Strip + Decongestant) | -1.69 (1.436)

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the investigational product and until 5 days following last administration of the investigational product.
Arm/Group | Marketed Nasal Strip | Placebo Nasal Strip | Decongestant | Marketed Nasal Strip Plus Decongestant
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.